CLINICAL TRIAL: NCT03384173
Title: Use of NIRS to Detect Acute Kidney Injury in Preterm Infants
Brief Title: NIRS Monitoring to Detect AKI in Preterm Infants
Acronym: nNIRS-AKI
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-0589; 2017-013 (Other: Meriter IRB); A536757 (Other: UW Madison); SMPH/PEDIATRICS/PEDIATRICS (Other: UW Madison)
Record Dates: First submitted 2017-12-15; First posted 2017-12-27 (Actual); Results first posted 2020-12-21 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-10

CONDITIONS: Acute Kidney Injury; Premature Infant
Keywords: Near Infrared Spectroscopy; Creatinine; Urine Output
MeSH Terms: conditions — Acute Kidney Injury; Premature Birth | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- NIRS monitoring: These infants will be monitored with NIRS
  Interventions: Device: Near Infrared Spectroscopy

INTERVENTIONS:
Device: Near Infrared Spectroscopy — Application of regional NIRS sensors to brain and kidney sites in the first 48 hours after birth to monitor regional tissue oxygenation for the first 7 days of age.
  Other Names: NIRS

SUMMARY:
This study will examine the relationship of oxygen levels, using Near-infrared spectroscopy (NIRS) monitoring, and kidney injury in infants born prematurely. NIRS is a skin sensor which detects the amount of oxygen going to different organs, most often used to monitor the brain and kidney.

DETAILED DESCRIPTION:
This prospective, single-center study was conducted at UnityPoint Health-Meriter Hospital (Madison, WI, USA) in preterm neonates admitted to a level III NICU from April 2018 to August 2019. The primary study aim was to assess changes in RrSO2 with continuous renal NIRS monitoring to detect AKI during the first 7 days of age.

The INVOS 5100 C (Somanetics, Troy, MI, USA) four channel NIRS monitors were used to measure RrSO2 (measured at the right or left flank) and Cerebral regional Somatic tissue Oxygenation (CrSO2; measured at the forehead) for all neonates. At each measurement site, for skin protection, subjects had a transparent Mepitel (with Safetac Technology, Norcross, GA) adhesive dressing placed with the adhesive neonatal NIRS sensor (INVOS OxyAlert NIRSensor, Covidien) adhered over the Mepitel dressing. Neither cerebral or kidney sensors were placed with ultrasound guidance. Tissue oxygenation was recorded every 3 seconds until 7 days of age, and the sensor was changed one time when the patient reached three to four days of age per the company's recommendation. There were no restrictions on positioning or handling of neonates; nurses re-positioned neonates every 3-6 hours per unit protocol to prevent skin pressure injuries. Researchers, staff, and parents were blinded to RrSO2 values.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants < 32 weeks
* Admitted to Unity Point Health(UPH) Meriter Newborn Intensive Care Unit (NICU)
* Application of NIRS by 48 hours of age

Exclusion Criteria:

* Congenital anomaly of the kidney or urinary tract (CAKUT)

Ages: 1 Minute to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants that are less than 32 weeks, admitted to Unity Point Health(UPH) Meriter Newborn Intensive Care Unit (NICU) with application of NIRS by 48 hours of age.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Harer, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UnityPoint Health Meriter Hospital, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chock VY, Rose LA, Mante JV, Punn R. Near-infrared spectroscopy for detection of a significant patent ductus arteriosus. Pediatr Res. 2016 Nov;80(5):675-680. doi: 10.1038/pr.2016.148. Epub 2016 Sep 7. PMID 27603562
- [Background] Ruf B, Bonelli V, Balling G, Horer J, Nagdyman N, Braun SL, Ewert P, Reiter K. Intraoperative renal near-infrared spectroscopy indicates developing acute kidney injury in infants undergoing cardiac surgery with cardiopulmonary bypass: a case-control study. Crit Care. 2015 Jan 29;19(1):27. doi: 10.1186/s13054-015-0760-9. PMID 25631390
- [Background] Hazle MA, Gajarski RJ, Aiyagari R, Yu S, Abraham A, Donohue J, Blatt NB. Urinary biomarkers and renal near-infrared spectroscopy predict intensive care unit outcomes after cardiac surgery in infants younger than 6 months of age. J Thorac Cardiovasc Surg. 2013 Oct;146(4):861-867.e1. doi: 10.1016/j.jtcvs.2012.12.012. Epub 2013 Jan 12. PMID 23317940
- [Background] Owens GE, King K, Gurney JG, Charpie JR. Low renal oximetry correlates with acute kidney injury after infant cardiac surgery. Pediatr Cardiol. 2011 Feb;32(2):183-8. doi: 10.1007/s00246-010-9839-x. Epub 2010 Nov 19. PMID 21085945
- [Background] McNeill S, Gatenby JC, McElroy S, Engelhardt B. Normal cerebral, renal and abdominal regional oxygen saturations using near-infrared spectroscopy in preterm infants. J Perinatol. 2011 Jan;31(1):51-7. doi: 10.1038/jp.2010.71. Epub 2010 Jun 10. PMID 20539273

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NIRS Monitoring
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- No Acute Kidney Injury (AKI): Infants with No AKI diagnosis.
  These infants will be monitored with NIRS
  Near Infrared Spectroscopy: Application of regional NIRS sensors to brain and kidney sites in the first 48 hours after birth to monitor regional tissue oxygenation for the first 7 days of age.
- Acute Kidney Injury (AKI): Infants diagnosed with AKI.
  These infants will be monitored with NIRS
  Near Infrared Spectroscopy: Application of regional NIRS sensors to brain and kidney sites in the first 48 hours after birth to monitor regional tissue oxygenation for the first 7 days of age.
- Total: Total of all reporting groups
Arm/Group | No Acute Kidney Injury (AKI) | Acute Kidney Injury (AKI) | Total
Number analyzed (Participants) | 32 | 3 | 35
Age, Continuous [Median (Inter-Quartile Range); unit: gestational age (weeks)] | 29.4 [26.9 to 30.6] | 25 [23 to 27.3] | 27.2 [23 to 30.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 3 | 16
  Male | 19 | 0 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 29 | 3 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 1 | 12
  White | 18 | 1 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 32 | 3 | 35
Small for gestational age [Number; unit: participants] — Small for gestational age defined as <10% for birthweight on the Fenton Growth Chart.
  participants | 3 | 2 | 5
Birth Weight [Median (Inter-Quartile Range); unit: grams] | 1135 [823 to 1490] | 655 [485 to 1020] | 945 [485 to 1490]

OUTCOME MEASURES:

1. Primary Outcome: Renal NIRS Tissue Oxygenation Differential
Description: Comparison of Renal saturation (Rsat) in neonates with AKI to those without AKI. RSO2 will be recorded until 7 days of age. Median RSO2 for 1 week and median for individual days 2-7 will be calculated.
  The INVOS 5100 C (Somanetics, Troy, MI, USA) four channel NIRS monitors will be used to measure renal regional oxygenation (RrSO2) values for all neonates.
Time Frame: Up to 1 week
Measure: Median (Inter-Quartile Range); unit: percentage saturation
Arm/Group | No Acute Kidney Injury (AKI) | Acute Kidney Injury (AKI)
Number analyzed (Participants) | 32 | 3
percentage saturation
  1 week Median RSO2 | 60 [58.4 to 62] | 32.4 [27.9 to 47.1]
  Day 2 RrSO2 | 62.5 [59 to 65.7] | 44.4 [39.4 to 46.6]
  Day 3 RrSO2 | 60.4 [59.3 to 61.7] | 30.8 [28 to 33]
  Day 4 RrSO2 | 59.1 [57 to 59.9] | 29.9 [27 to 31.7]
  Day 5 RrSO2 | 59.7 [58.4 to 61.1] | 29.2 [25.7 to 36.9]
  Day 6 RrSO2 | 60 [59 to 61.3] | 24 [20.9 to 27.8]
  Day 7 RrSO2 | 60.3 [57.8 to 66.9] | 55.3 [39 to 58.7]
Statistical Analysis 1: Comparison: No Acute Kidney Injury (AKI) vs Acute Kidney Injury (AKI); Test type: Superiority; p < 0.001, ANOVA

2. Secondary Outcome: Correlation of Renal NIRS Values to Serum Creatinine
Description: At each time a serum creatinine was collected, the RrSO2 value was recorded.
Time Frame: Days 1-7 of age
Population: All participants with serum creatinine values were included
Measure: Median (Inter-Quartile Range); unit: mg/dL
Groups:
- Infants With Serum Creatinine Values: Any infant with serum creatinine values were included.
Arm/Group | Infants With Serum Creatinine Values
Number analyzed (Participants) | 35
mg/dL | 0.81 [0.67 to 0.93]
Statistical Analysis 1: Comparison: Infants With Serum Creatinine Values; Test type: Other — Correlation, Pearson r; p = 0.17, Pearson r correlation; Pearson r correlation = 0.16, 95% CI 2-sided [-0.07 to 0.37]

3. Secondary Outcome: Correlation of Renal NIRS Values to Urine Output
Description: In patients with urine output recorded, it was compared to RrSO2 values
Time Frame: Days 1-7 of age
Population: All patients
Measure: Median (Inter-Quartile Range); unit: mL/kg/hour
Groups:
- Neonates With Urine Output Recorded: All neonates with urine output recorded were included
Arm/Group | Neonates With Urine Output Recorded
Number analyzed (Participants) | 35
mL/kg/hour | 3 [2.3 to 4.5]
Statistical Analysis 1: Comparison: Neonates With Urine Output Recorded; Test type: Other — Correlation, Pearson r; p = 0.32, Pearson r correlation; Pearson r correlation = 0.12, 95% CI 2-sided [-0.11 to 0.33]

4. Secondary Outcome: Baseline Renal NIRS Values Before Caffeine
Description: these are the average renal NIRS values over 6 hours prior to a dose of caffeine broken down by percentage
Time Frame: Baseline (6 hours prior to caffeine dose)
Population: Out of 35 enrolled participants, 32 participants received total 156 doses of caffeine. Giving Caffeine was at the discretion of the attending physician.
  This analysis is done by the dose of caffeine, and not the participant. Each row shows the number of doses given in that baseline percentage.
  The caffeine doses have been de-identified from the participants so the number of participants in each row cannot be calculated from the currently recorded data.
Measure: Median (Inter-Quartile Range); unit: % oxygenation
Units Other Than Participants: caffeine doses
Groups:
- Baseline Renal NIRS Values Before Caffeine: 6 hour average prior to dose of caffeine
Arm/Group | Baseline Renal NIRS Values Before Caffeine
Number analyzed (Participants) | 32
Number analyzed (caffeine doses) | 156
% oxygenation
  Baseline <20% (12 caffeine doses): number analyzed (caffeine doses) | 12
  Baseline <20% (12 caffeine doses) | 15.24 [15.01 to 16.86]
  Baseline 20-29.99% (16 caffeine doses): number analyzed (caffeine doses) | 16
  Baseline 20-29.99% (16 caffeine doses) | 26.93 [22.25 to 28.83]
  Baseline 30-39.99% (18 caffeine doses): number analyzed (caffeine doses) | 18
  Baseline 30-39.99% (18 caffeine doses) | 36.11 [34.13 to 38.8]
  Baseline 40-49.99% (13 caffeine doses): number analyzed (caffeine doses) | 13
  Baseline 40-49.99% (13 caffeine doses) | 48.61 [43.65 to 49.4]
  Baseline 50-59.99% (21 caffeine doses): number analyzed (caffeine doses) | 21
  Baseline 50-59.99% (21 caffeine doses) | 54.41 [51.78 to 57.33]
  Baseline >60% (76 caffeine doses): number analyzed (caffeine doses) | 76
  Baseline >60% (76 caffeine doses) | 73.08 [66.82 to 80.49]

5. Secondary Outcome: Renal NIRS Values 1 Hour After Caffeine
Description: Renal NIRS values one hour after caffeine broken down by baseline average.
Time Frame: At 1 hour after caffeine dose
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percentage saturation
Units Other Than Participants: caffeine doses
Arm/Group | NIRS Monitoring
Number analyzed (Participants) | 32
Number analyzed (caffeine doses) | 156
percentage saturation
  Doses with baseline <20% (12 caffeine doses): number analyzed (caffeine doses) | 12
  Doses with baseline <20% (12 caffeine doses) | 16.09 [15.1 to 17.45]
  Doses with baseline 20-29.99% (16 caffeine doses): number analyzed (caffeine doses) | 16
  Doses with baseline 20-29.99% (16 caffeine doses) | 32.83 [26.38 to 38.6]
  Doses with baseline 30-39.99% (18 caffeine doses): number analyzed (caffeine doses) | 18
  Doses with baseline 30-39.99% (18 caffeine doses) | 44.18 [34.65 to 51.26]
  Doses with baseline 40-49.99% (13 caffeine doses): number analyzed (caffeine doses) | 13
  Doses with baseline 40-49.99% (13 caffeine doses) | 49.23 [45.71 to 55.01]
  Doses with baseline 50-59.99% (21 caffeine doses): number analyzed (caffeine doses) | 21
  Doses with baseline 50-59.99% (21 caffeine doses) | 54.31 [51.51 to 60.61]
  Doses with baseline >60% (76 caffeine doses): number analyzed (caffeine doses) | 76
  Doses with baseline >60% (76 caffeine doses) | 70.55 [63.44 to 77.55]
Statistical Analysis 1: Comparison: NIRS Monitoring; Control group is Secondary analysis #4, baseline values before caffeine dose; Test type: Other — Mann Whitney U non parametric test; p < 0.01, Wilcoxon (Mann-Whitney) — A-priori threshold p<0.05 for 'subgroup 20-29.99%' vs 'baseline value before caffeine dose'. A-priori threshold p<0.05 for 'subgroup 30-39.99%' vs 'baseline value before caffeine dose'

6. Secondary Outcome: Renal NIRS Values 2 Hours After Caffeine
Description: Renal NIRS values 2 hours after caffeine broken down by baseline average
Time Frame: At 2 hours after caffeine dose
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percentage saturation
Units Other Than Participants: caffeine doses
Arm/Group | NIRS Monitoring
Number analyzed (Participants) | 32
Number analyzed (caffeine doses) | 156
percentage saturation
  Doses with baseline <20% (12 caffeine doses): number analyzed (caffeine doses) | 12
  Doses with baseline <20% (12 caffeine doses) | 16.15 [15.11 to 21.61]
  Doses with baseline 20-29.99% (16 caffeine doses): number analyzed (caffeine doses) | 16
  Doses with baseline 20-29.99% (16 caffeine doses) | 40.66 [32.83 to 47.75]
  Doses with baseline 30-39.99% (18 caffeine doses): number analyzed (caffeine doses) | 18
  Doses with baseline 30-39.99% (18 caffeine doses) | 39.06 [26.85 to 49.9]
  Doses with baseline 40-49.99% (13 caffeine doses): number analyzed (caffeine doses) | 13
  Doses with baseline 40-49.99% (13 caffeine doses) | 49.96 [43.6 to 56.03]
  Doses with baseline 50-59.99% (21 caffeine doses): number analyzed (caffeine doses) | 21
  Doses with baseline 50-59.99% (21 caffeine doses) | 55.81 [49.06 to 63.2]
  Doses with baseline >60% (76 caffeine doses): number analyzed (caffeine doses) | 76
  Doses with baseline >60% (76 caffeine doses) | 68.51 [62.63 to 78.68]
Statistical Analysis 1: Comparison: NIRS Monitoring; Control group is secondary outcome #4, baseline values before caffeine dose; Test type: Other — Mann Whitney U non parametric test; p < 0.001, Wilcoxon (Mann-Whitney) — A-priori threshold p<0.05 for 'subgroup 20-29.99%' vs 'baseline value before caffeine dose'

7. Secondary Outcome: Renal NIRS Values 3 Hours After Caffeine
Description: Renal NIRS values 3 hours after caffeine broken down by baseline average
Time Frame: At 3 hours after caffeine dose
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percentage saturation
Units Other Than Participants: caffeine doses
Arm/Group | NIRS Monitoring
Number analyzed (Participants) | 32
Number analyzed (caffeine doses) | 156
percentage saturation
  Doses with baseline <20% (12 caffeine doses): number analyzed (caffeine doses) | 12
  Doses with baseline <20% (12 caffeine doses) | 17.3 [16.09 to 30.97]
  Doses with baseline 20-29.99% (16 caffeine doses): number analyzed (caffeine doses) | 16
  Doses with baseline 20-29.99% (16 caffeine doses) | 36.12 [33.25 to 41.48]
  Doses with baseline 30-39.99% (18 caffeine doses): number analyzed (caffeine doses) | 18
  Doses with baseline 30-39.99% (18 caffeine doses) | 40.4 [30.55 to 51.71]
  Doses with baseline 40-49.99% (13 caffeine doses): number analyzed (caffeine doses) | 13
  Doses with baseline 40-49.99% (13 caffeine doses) | 50.6 [47.21 to 54.98]
  Doses with baseline 50-59.99% (21 caffeine doses): number analyzed (caffeine doses) | 21
  Doses with baseline 50-59.99% (21 caffeine doses) | 58.05 [53.22 to 63.53]
  Doses with baseline >60% (76 caffeine doses): number analyzed (caffeine doses) | 76
  Doses with baseline >60% (76 caffeine doses) | 66.55 [61.92 to 74.7]
Statistical Analysis 1: Comparison: NIRS Monitoring; Comparison group is Secondary outcome #4, baseline caffeine values by subgroup; Test type: Other — Mann-Whitney U non parametric t test; p < 0.01, Wilcoxon (Mann-Whitney) — A-priori threshold p<0.05 for 'subgroup 20-29.99%' vs 'baseline value before caffeine dose'. A-priori threshold p<0.05 for 'subgroup >60% ' vs 'baseline value before caffeine dose'

8. Secondary Outcome: Renal NIRS Values 4 Hours After Caffeine
Description: Renal NIRS values 4 hours after caffeine broken down by baseline average
Time Frame: At 4 hours after caffeine dose
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percentage saturation
Units Other Than Participants: caffeine doses
Arm/Group | NIRS Monitoring
Number analyzed (Participants) | 32
Number analyzed (caffeine doses) | 156
percentage saturation
  Doses with baseline <20% (12 caffeine doses): number analyzed (caffeine doses) | 12
  Doses with baseline <20% (12 caffeine doses) | 16.98 [15.01 to 22.93]
  Doses with baseline 20-29.99% (16 caffeine doses): number analyzed (caffeine doses) | 16
  Doses with baseline 20-29.99% (16 caffeine doses) | 39.64 [33.55 to 48.35]
  Doses with baseline 30-39.99% (18 caffeine doses): number analyzed (caffeine doses) | 18
  Doses with baseline 30-39.99% (18 caffeine doses) | 42.71 [29.96 to 54.29]
  Doses with baseline 40-49.99% (13 caffeine doses): number analyzed (caffeine doses) | 13
  Doses with baseline 40-49.99% (13 caffeine doses) | 48.47 [45.52 to 53.01]
  Doses with baseline 50-59.99% (21 caffeine doses): number analyzed (caffeine doses) | 21
  Doses with baseline 50-59.99% (21 caffeine doses) | 57.78 [52.05 to 64.33]
  Doses with baseline >60% (76 caffeine doses): number analyzed (caffeine doses) | 76
  Doses with baseline >60% (76 caffeine doses) | 71.19 [62.12 to 79.68]
Statistical Analysis 1: Comparison: NIRS Monitoring; Comparison group is secondary outcome #4, baseline values before caffeine dose; Test type: Other; p < 0.0001, Wilcoxon (Mann-Whitney) — A-priori threshold p<0.05 for 'subgroup 20-29.99%' vs 'baseline value before caffeine dose'

9. Secondary Outcome: Renal NIRS Values 6 Hours After Caffeine
Description: Renal NIRS values 6 hours after caffeine broken down by baseline average
Time Frame: At 6 hours after caffeine dose
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percentage saturation
Units Other Than Participants: caffeine doses
Arm/Group | NIRS Monitoring
Number analyzed (Participants) | 32
Number analyzed (caffeine doses) | 156
percentage saturation
  Doses with baseline <20% (12 caffeine doses): number analyzed (caffeine doses) | 12
  Doses with baseline <20% (12 caffeine doses) | 15.4 [15.03 to 23.82]
  Doses with baseline 20-29.99% (16 caffeine doses): number analyzed (caffeine doses) | 16
  Doses with baseline 20-29.99% (16 caffeine doses) | 35.18 [24.22 to 43.08]
  Doses with baseline 30-39.99% (18 caffeine doses): number analyzed (caffeine doses) | 18
  Doses with baseline 30-39.99% (18 caffeine doses) | 40.62 [33.47 to 51.59]
  Doses with baseline 40-49.99% (13 caffeine doses): number analyzed (caffeine doses) | 13
  Doses with baseline 40-49.99% (13 caffeine doses) | 49.97 [44.94 to 57.21]
  Doses with baseline 50-59.99% (21 caffeine doses): number analyzed (caffeine doses) | 21
  Doses with baseline 50-59.99% (21 caffeine doses) | 55.8 [43.07 to 65.74]
  Doses with baseline >60% (76 caffeine doses): number analyzed (caffeine doses) | 76
  Doses with baseline >60% (76 caffeine doses) | 70.09 [62.65 to 79.39]
Statistical Analysis 1: Comparison: NIRS Monitoring; Comparison group is Secondary Outcome #4, baseline before dose of caffeine; Test type: Other — Mann Whitney U non-parametric t-test; p < 0.05, Wilcoxon (Mann-Whitney) — A-priori threshold p<0.05 for 'subgroup 20-29.99%' vs 'baseline value before caffeine dose'

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | No Acute Kidney Injury (AKI) | Acute Kidney Injury (AKI)
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/3
Other Adverse Events (participants affected / at risk) | 0/32 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT03384173/Prot_SAP_000.pdf